CLINICAL TRIAL: NCT03204253
Title: Effects of Recombinant LH in Late Phase of Ovarian Stimulation in Patients With Repeated Implantation Failure, Clinical Results
Brief Title: Effects of Recombinant LH in Patients With Repeated Implantation Failure
Acronym: late-rLH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Davide Francomano, PHD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Biofertility
Record Dates: First submitted 2016-12-09; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Female Infertility; Female Subfertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rFSH + r-LH in combination (Experimental): treatment group
  Interventions: Drug: rFSH + r-LH in combination
- rFSH alone (Active Comparator): control group
  Interventions: Drug: rFSH alone

INTERVENTIONS:
Drug: rFSH + r-LH in combination — 29 women stimulated with rFSH supplemented by rLH in the late follicular phase started at the same time of starting the antagonist administration.
  Arms: rFSH + r-LH in combination
Drug: rFSH alone — 32 women who were stimulated with recombinant FSH alone
  Arms: rFSH alone

SUMMARY:
Pregnancy rates fall dramatically in women after 35 years undergoing to IVF or ICSI. While ovarian aging obviously plays the major role in this phenomenon, over suppression of endogenous LH concentrations with GnRH agonists or antagonists-an integral part of standard IVF/ ICSI protocols-may also play a pivotal role.

Assisted reproduction technology protocols using GnRH agonists have been considered as the standard protocol during the last two decades, but the use of GnRH antagonists offers the opportunity to control the endogenous LH surge in a rapid and more convenient way.

LH plays a key role in the intermediate-late phases of folliculogenesis. The presence of receptors for LH in cumulus granulosa cells and its correlation with oocyte maturation has been demonstrated. Although ovarian stimulation is efficiently achieved in most cases by the administration of exogenous FSH alone, specific subgroups of women may benefit from LH activity supplementation during ovarian stimulation. Some authors have found improved outcome with LH activity supplementation in advanced reproductive age women.

LH has a number of roles in follicular development, induction of ovulation, completion of meiosis I, early luteinization and the production of progesterone.

The efficacy of recombinant human follicle-stimulating hormone (r-hFSH) for ovarian stimulation is well established however, the role of supplementary recombinant human luteinizing hormone (r-hLH) is less clear.

Aim of the present study is to evaluate If adding rLH in the late phase of stimulation can benefit in some patient awith repeated implantation failure.

DETAILED DESCRIPTION:
Study Design, Size and Duration

The study was conducted at the - Bio fertility IVF Center, Rome, Italy, on infertile couples due to male factor undergoing ICSI treatment.

The study was reviewed and approved by the institutional review board at the - Biofertilty IVF Center.

All patients undergoing ICSI and participating in the study gave informed consent.

Patients included in the study had regular spontaneous menstrual cycles (26-39 days) and were aged < 42 years.

All patients had acceptable follicular phase serum concentrations of FSH (≤10IU/L), LH (<10IU/L) and oestradiol (<60pg/ml), body mass index (BMI) ≤ 30 kg/m2, presence of both ovaries and normal uterine cavity.

Only patients with repeated implantation failure in at least two previous IVF cycles were included.

Patients were excluded from the study if they had any clinically significant systemic disease, polycystic ovarian syndrome (PCOS), a previous history of severe ovarian hyperstimulation syndrome (OHSS), abnormal gynaecological bleeding of unknown origin, a previous history of intolerance to any of the agents used in the study.

This was a prospective, randomized study.

All patient sighed a detailed informed consent.

The study is in accordance to the GCP guidelines

They were randomly divided into two groups (A and B).

All patients were stimulated in GnRH antagonist flexible protocol cycles using rFSH started on day 2 of a spontaneous or induced cycle. HCG (10000 iu ) was administered by I.M route when at least 2 folliclesreached 18 mm in diameter.

Group A included 29 women stimulated with rFSH supplemented by rLH in the late follicular phase started at the same time of starting the antagonist administration.

Those patients received 75 iu of rLH (Luveris serono) daily and 150 iu about 12 hours before triggering ovulation with HCG while Group B included 32 women who were stimulated with recombinant FSH (gonal F serono) only. The oocytes were decumulated and assessed for the maturation two hours after pick up which was done 36 hours after hcg injection. Mature oocyte should have an intact first polar body and homogeneously fine granular and light-colored ooplasm

The rate of metaphase II oocytes was calculated and the MII oocytes were assessed for cytoplasmic morphology and maturity. MII oocytes with a light color and fine homogeneous granulate ooplasm were considered oocytes normal morphology and classified as oocytes that have completed their cytoplasmic maturation.

Embryo transfer was done after 2 days of icsi. Pregnancy test was done after 12 days and clinical pregnancy and number of gestional sacs were assured after 2 weeks of positive pregnancy test with presence of featal heart beats. The mean, SD, T-test and Chi square test were used for statistic calculations of the results.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with repeated implantation failure in at least two previous IVF cycles were included.

Exclusion Criteria:

* Patients were excluded from the study if they had any clinically significant systemic disease, polycystic ovarian syndrome (PCOS), a previous history of severe ovarian hyperstimulation syndrome (OHSS), abnormal gynaecological bleeding of unknown origin, a previous history of intolerance to any of the agents used in the study.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of ovocites retrived | 1 cicle of stimulation of 14 days
  Possible beneficial effects of rLH in the late phase of stimulation in patient with repeated implantation failure

CONTACTS AND LOCATIONS:
Overall Officials: Davide Francomano, Principal Investigator — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: No